CLINICAL TRIAL: NCT03218085
Title: Role of Exogenous and Endogenous Sex Hormones on Tenofovir and Emtricitabine
Brief Title: Role of Exogenous and Endogenous Sex Hormones on Tenofovir and Emtricitabine Disposition in Female Genital Tract
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Sponsor
Other Study IDs: PHARM-2016-24820
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: HIV/AIDS; Menopause; Inflammation Vagina
Keywords: tenofovir; prevention; microbiome; cervicovaginal; biopsy; swab; cytokines; inflammation; pharmacology
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Vaginitis; Inflammation | interventions — Tenofovir; Emtricitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tenofovir — Two cervical biopsies, blood plasma, PBMC, and two cervicovaginal swabs will be collected at a single study visit
Drug: Emtricitabine — Two cervical biopsies, blood plasma, PBMC, and two cervicovaginal swabs will be collected at a single study visit

SUMMARY:
Cervical biopsies will be collected from women aged 18 and over whom are virally suppressed and taking tenofovir as part of their antiretroviral therapy regimen. Blood plasma, peripheral blood mononuclear cells (PBMC), and cervicovaginal swabs will also be collected. Drug concentrations, hormone concentrations, inflammatory cytokines, and vaginal microbiome will be evaluated to understand the role of hormones, inflammation, and the microbiome in modulating drug efficacy in the female genital tract.

ELIGIBILITY:
Inclusion Criteria:

1. Female, or transgender female with a cervix, age 18 years or older
2. HIV-positive
3. Stable on antiretroviral regimen containing tenofovir or emtricitabine for at least 2 weeks at time of enrollment.
4. Virally suppressed (HIV-RNA copies <50 copies/mL) for at least 6 months at time of enrollment.
5. Willing to refrain from vaginal intercourse and use of vaginal devices such as douches and sex toys within 72 hours of the biopsy visit.
6. Willing and able to give signed informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Currently pregnant or previous pregnancy within 3 months of enrollment
  2. Currently breast feeding
  3. Symptomatic vaginal infection within 2 weeks prior to enrollment
  4. Unexplained, undiagnosed abnormal bleeding per vagina, bleeding per vagina during or following vaginal intercourse, or gynecologic surgery within 90 days prior to enrollment
  5. Use of oral and/or vaginal preparations of antibiotic or antifungal medications within 30 days prior to the enrollment visit
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Assess the influence of exogenous and endogenous sex hormones on tenofovir and emtricitabine concentrations in cervical tissues | Day 1

SECONDARY OUTCOMES:
To assess the influence of endogenous and exogenous sex hormones on the expression of drug metabolizing enzymes and transporters in cervical tissue | Day 1
To determine the influence of endogenous and exogenous sex hormones on the endogenous nucleotide pool in cervical tissues | Day 1
To discriminate between local and systemic effects of hormonal use on antiretroviral disposition. | Day 1
To determine relationship between local inflammation and drug disposition in the female genital tract | Day 1
To identify potential role of the vaginal microbiome in local drug disposition, | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States